CLINICAL TRIAL: NCT03590561
Title: Einfluss Von Hochkalorischer Nahrungsaufnahme Auf Die Insulinsensitivität Des Menschlichen Zentralnervensystems
Brief Title: Effect of High Caloric Diet on Brain Insulin Sensitivity and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 813/2017BO2
Record Dates: First submitted 2018-06-14; First posted 2018-07-18 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High caloric diet (Experimental): Participants will eat 1500 kcal more than their usual diet for five days.
  Interventions: Other: High caloric diet
- Control diet (No Intervention): Participants will eat regular diet.

INTERVENTIONS:
Other: High caloric diet — After dietary counseling, subjects will receive high caloric snacks for five days.
  Arms: High caloric diet

SUMMARY:
Obesity if known to be associated with brain insulin resistance in humans and evidence is rapidly accumulating that brain insulin resistance influences peripheral metabolism, eating behavior and cognition. A reduced insulin response in the brain is found mainly in people with a metabolically unfavorable fat distribution - high visceral fat. Visceral fat produces inflammatory mediators and elevated inflammatory levels are closely linked to insulin resistance. Inflammation of the brain (i.e., neuroinflammation) has been proposed as a possible cause of brain insulin resistance. Interestingly, rodent models of a high calorie diet show that these inflammatory mechanisms occur rapidly in the brain, even prior to weight gain of the animals. Among other things, it has been shown in humans that a short-term increase in calories, especially carbohydrates and fats, reduces insulin sensitivity in the body and increases inflammatory parameters in the blood. Whether a high-calorie diet triggers insulin resistance or inflammation in the human brain is currently unknown.

Aim of study:

The aim of the study is to investigate the effects of a five-day high calorie diet in healthy young male volunteers on peripheral and brain insulin sensitivity as well as on eating behavior, mood and cognition. Brain insulin sensitivity, peripheral metabolism and different behavioral assessments will be evaluated before, 1 week and 2 weeks after high caloric diet.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-24 kg/m2

  * Non smoking
  * normal glucose tolerance during 75g oral glucose tolerance test (OGTT)
  * Exercise less than 2h per week

Exclusion Criteria:

* Vegetarians and Vegans
* Food allergies
* Working at night
* Professional Athletes
* Not removable metal parts in or on the body
* manifest cardiovascular disease
* claustrophobia
* recent surgery (less than 3 months)
* Simultaneous participation in other studies
* Acute disease or infection within the last 4 weeks
* neurological and psychiatric disorders
* treatment with centrally acting drugs
* hemoglobin Hb <13g / dl
* Hypersensitivity to any of the substances used

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change in brain insulin sensitivity | Outcome measurements will be assessed at baseline (t0). Then, the 5-day high caloric diet or control dietwill start 5 to 30 days after t0. Outcome measurements will again be assessed on the 6th-7th day and on the 10th-15th day after start of diet.
  fMRI measurement will be performed before and after administration of 160 U of human insulin as nasal spray. Changes in regional activity will be quantified to assess regional brain insulin sensitivity.
Change in quantitative proton density | Outcome measurements will be assessed at baseline (t0). Then, the 5-day high caloric diet or control dietwill start 5 to 30 days after t0. Outcome measurements will again be assessed on the 6th-7th day and on the 10th-15th day after start of diet.
  The inflammatory processes in the brain will be measured through the quantification of the water content by means of proton density imaging.
Change in brain metabolites | Outcome measurements will be assessed at baseline (t0). Then, the 5-day high caloric diet or control dietwill start 5 to 30 days after t0. Outcome measurements will again be assessed on the 6th-7th day and on the 10th-15th day after start of diet.
  The inflammatory processes in the brain will be measured through the determination of brain metabolites by MR spectroscopy

SECONDARY OUTCOMES:
Change in whole-body insulin sensitivity | Outcome measurements will be assessed at baseline (t0). Then, the 5-day high caloric diet or control diet will start 5 to 30 days after t0. Outcome measurements will again be assessed on the 6th-7th day and on the 10th-15th day after start of diet.
  Insulin sensitivity will be estimated from a frequent-sampling 75 g oral glucose tolerance test using the Matsuda formula.
Change in body fat distribution | Outcome measurements will be assessed at baseline (t0). Then, the 5-day high caloric diet or control dietwill start 5 to 30 days after t0. Outcome measurements will again be assessed on the 6th-7th day and on the 10th-15th day after start of diet.
  Body composition will be addressed by whole-body MRI and liver MRS.
Behavioral assessment | Outcome measurements will be assessed at baseline (t0). Then, the 5-day high caloric diet or control dietwill start 5 to 30 days after t0. Outcome measurements will again be assessed on the 6th-7th day and on the 10th-15th day after start of diet.
  Memory function, food reward behavior and mood will be assessed by questionnaires, neuropsychological testing and a snack test.
Change in insulin secretion | Outcome measurements will be assessed at baseline (t0). Then, the 5-day high caloric diet or control dietwill start 5 to 30 days after t0. Outcome measurements will again be assessed on the 6th-7th day and on the 10th-15th day after start of diet.
  Insulin secretion will be estimated from a frequent-sampling 75 g oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
We will not able to share individual participant data due to data protection restraints.